CLINICAL TRIAL: NCT03482115
Title: Whole Brain Connectivity Changes Induced by Traumatic Coma: Combined Structural, Functional and Neuroinflammatory Approaches
Brief Title: Brain Network Disruptions Related to Traumatic Coma
Acronym: Coma3D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/16/8257; 2017-001986-26 (EudraCT Number)
Record Dates: First submitted 2018-02-08; First posted 2018-03-29 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Traumatic Coma
Keywords: coma; traumatic brain injury; anoxic encephalopathy; brain connectome; neuroinflammation; prognosis
MeSH Terms: conditions — Coma, Post-Head Injury; Coma; Brain Injuries, Traumatic; Hypoxia, Brain; Neuroinflammatory Diseases | interventions — N,N-diethyl-2-(2-(4-(2-fluoroethoxy)phenyl)-5,7-dimethylpyrazolo(1,5-a)pyrimidin-3-yl)acetamide; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comatose patient (Experimental): Subject with coma of traumatic or anoxic aetiology : PET examination with radiopharmaceutical drug [18F] DPA-714, MRI examination and Blood samples.
  Interventions: Radiation: PET examination with radiopharmaceutical drug [18F] DPA-714; Diagnostic Test: MRI examination; Biological: Blood samples
- control volunteers (Other): subject control : PET examination with radiopharmaceutical drug [18F] DPA-714, MRI examination and Blood samples.
  Interventions: Radiation: PET examination with radiopharmaceutical drug [18F] DPA-714; Diagnostic Test: MRI examination; Biological: Blood samples

INTERVENTIONS:
Radiation: PET examination with radiopharmaceutical drug [18F] DPA-714 — Using a Biograph 6 Truepoint device. Establishment of a venous route. It will be injected 4 MBq / kg of 18F-DPA714 by the venous route with a maximum dose of 280 MBq. The patient will be placed along the orbito-meatal line. Brain acquisition will begin 60 minutes post-injection
Diagnostic Test: MRI examination — MRI device Philips Achieva - 3Tesla. The acquisition of the data will include different sequences (anatomical MRI, diffusion MRI, resting fMRI) and will last a total of one hour (installation and removal of the patient in the machine included).anatomical MRI associated with FLAIR (Fluid Attenuation Inversion Recovery) and diffusion tensor (tractography).
Biological: Blood samples — Characterization of the TSPO phenotype (mitochondrial translocase) for tracer affinity

SUMMARY:
To provide a fine-grained description of the brain network dysfunctions induced by severe traumatic brain injury (TBI) or anoxic encephalopathy, that are responsible for the acute state of unarousable unawareness, named coma, this trial wants to explore the usefulness in this setting of a combined neuroimaging approaches encompassing several up-to-date techniques as structural MRI, fMRI and positron emission tomography (PET) scan (neuroinflammation ligands).

DETAILED DESCRIPTION:
So far, the gold standard for neuroprognostication of severe traumatic brain injury (TBI) or anoxic encephalopathy is the bedside behavioural evaluation. Nevertheless, the predictive value of such an exclusive clinical approach has been consistently reported as limited and insufficient in this challenging clinical setting. Recent theoretical and experimental data converge towards the idea of the critical implication of long-range brain connection in consciousness access and maintain. Nevertheless, previous studies have focused on the specific analysis of some targeted connections (regions of interest), and have used exclusively a single approach in neuroimaging (structural or functional imaging), with no interest in the neuro-inflammatory and neurodegenerative mechanisms likely associated with these disconnection phenomena. So, cerebral disconnection characterization at the level of the whole brain, at different stages of pathological abolition of consciousness must be made, on an anatomical, functional and metabolic scale. This descriptive study represents a first step in the identification of relevant multimodal imaging biomarkers. This will then lead to a larger study to identify the prognostic impact of these different biomarkers obtained in the acute phase of patient management.

ELIGIBILITY:
Inclusion criteria for patients:

* Male or female / age between 18 to 75 years.
* Coma of traumatic or anoxic aetiology (GCS < 10).
* Early (< 1 month after TBI) and after the complete withdrawal of sedative agents.
* Written agreement for participation (legal responsible).

Inclusion criteria for controls:

* Male or female / age between 18 to 75 years, paired with patients (gender and age).
* Written agreement for participation

Exclusion criteria:

* Patients without public insurance regime.
* Pregnancy.
* Specific contraindication to the use of MRI (metallic material) or PET (specific allergy related to the ligand).

Exclusion criteria for controls:

- pharmacological treatments which could interfere with consciousness (left to the judgement of the investigator)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2021-11-07 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
Matrix of the neuroimaging data in PET examination | First Visit, within three days after day 0
  neuroinflammation by [18F] DPA-714 during PET imaging

SECONDARY OUTCOMES:
Glasgow Coma Scale (GCS) | Inclusion
  The Glasgow Coma Scale is divided into three components : ocular response (assessment 1-4 points), motor response (assessment 1-6 points) verbal response (evaluation of 1-5 points).
  Scores for each component are added together to get the total that will range between a minimum of 3 points (which corresponds to a patient who does not open his eyes and no motor response to stimulation or verbal response) and a maximum value of 15 points (corresponding to a patient with open eyes, obeying orders and maintaining a consistent language).
  It has been considered that the GCS score between 15 and 13 points corresponds to a slight alteration of consciousness, a score of 12-9 points with moderate impairment and 8 points or less with a serious deterioration in level of consciousness.
Coma Recovery Scale Revised (CRS-R) | 3 months +/- 3 days after the primary brain insult
  The Coma Recovery Scale Revised is divided into three components : return to consciousness (RECUP), vegetative neurological state (ENV) or minimal state of consciousness (ECM).
  This scale has been validated in French, with a value of Cronbach's Alpha estimated at 0.8.
  It is a score whose values are between 100 (normal level of consciousness) and 10 (coma). ENV and ECM have intermediate values (approximately 30 and 60, respectively).
FOUR score | 3 months +/- 3 days after the primary brain insult
  The FOUR score is a scale of 4 items and 16 points concerning qualitative behavioural assessment
analysis of imaging parameters obtained in MRI | First Visit, within three days after day 0
  assessing the strength of connectivity between different regions for the whole brain, measurement of anatomical connectivity, measurement of cortical thickness. All this measure use voxel/volume unit of the brain

CONTACTS AND LOCATIONS:
Overall Officials: Stein SILVA, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laureys S, Owen AM, Schiff ND. Brain function in coma, vegetative state, and related disorders. Lancet Neurol. 2004 Sep;3(9):537-46. doi: 10.1016/S1474-4422(04)00852-X. PMID 15324722
- [Background] Schiff ND. Recovery of consciousness after brain injury: a mesocircuit hypothesis. Trends Neurosci. 2010 Jan;33(1):1-9. doi: 10.1016/j.tins.2009.11.002. Epub 2009 Dec 1. PMID 19954851
- [Background] Silva S, de Pasquale F, Vuillaume C, Riu B, Loubinoux I, Geeraerts T, Seguin T, Bounes V, Fourcade O, Demonet JF, Peran P. Disruption of posteromedial large-scale neural communication predicts recovery from coma. Neurology. 2015 Dec 8;85(23):2036-44. doi: 10.1212/WNL.0000000000002196. Epub 2015 Nov 11. PMID 26561296
- [Background] Chauveau F, Van Camp N, Dolle F, Kuhnast B, Hinnen F, Damont A, Boutin H, James M, Kassiou M, Tavitian B. Comparative evaluation of the translocator protein radioligands 11C-DPA-713, 18F-DPA-714, and 11C-PK11195 in a rat model of acute neuroinflammation. J Nucl Med. 2009 Mar;50(3):468-76. doi: 10.2967/jnumed.108.058669. Epub 2009 Feb 17. PMID 19223401
- [Background] Arlicot N, Vercouillie J, Ribeiro MJ, Tauber C, Venel Y, Baulieu JL, Maia S, Corcia P, Stabin MG, Reynolds A, Kassiou M, Guilloteau D. Initial evaluation in healthy humans of [18F]DPA-714, a potential PET biomarker for neuroinflammation. Nucl Med Biol. 2012 May;39(4):570-8. doi: 10.1016/j.nucmedbio.2011.10.012. Epub 2011 Dec 14. PMID 22172392
- [Result] Sarton B, Tauber C, Fridman E, Peran P, Riu B, Vinour H, David A, Geeraerts T, Bounes F, Minville V, Delmas C, Salabert AS, Albucher JF, Bataille B, Olivot JM, Cariou A, Naccache L, Payoux P, Schiff N, Silva S. Neuroimmune activation is associated with neurological outcome in anoxic and traumatic coma. Brain. 2024 Apr 4;147(4):1321-1330. doi: 10.1093/brain/awae045. PMID 38412555
- [Derived] Mattia GM, Sarton B, Villain E, Vinour H, Ferre F, Buffieres W, Le Lann MV, Franceries X, Peran P, Silva S. Multimodal MRI-Based Whole-Brain Assessment in Patients In Anoxoischemic Coma by Using 3D Convolutional Neural Networks. Neurocrit Care. 2022 Aug;37(Suppl 2):303-312. doi: 10.1007/s12028-022-01525-z. Epub 2022 Jul 25. PMID 35876960